CLINICAL TRIAL: NCT02764437
Title: AsthMatic Inflammation and Neurocircuitry Activation (MINA)
Acronym: MINA
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-0021; 1R01HL123284-01A1 (NIH); A534220 (Other: UW Madison); SMPH\MEDICINE\ALLRGY&IMM (Other: UW Madison)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI-Bronch, PET-WLAC (Stress vs Control): Subjects will have a functional MRI scan 24 hours before a bronchoscopy with segmental allergen challenge. 48 hours post segmental allergen challenge, the subject will have another MRI and bronchoscopy. 4-6 weeks later, subjects will have a PET scan and whole lung antigen challenge under a stress condition or control condition. 4-6 weeks later, subject will have another PET scan and whole lung antigen challenge under a stress condition or control condition (whatever they did not have the first time).
  Interventions: Biological: Whole lung antigen challenge, segmental allergen challenge

INTERVENTIONS:
Biological: Whole lung antigen challenge, segmental allergen challenge — Whole lung antigen challenge with housedust mite, short ragweed or cat hair allergen extracts. Segmental allergen challenge with housedust mite, short ragweed or cat hair allergen extracts.
  Other Names: House dust mite, short ragweed, cat hair allergen extracts

SUMMARY:
The investigators have identified areas of the brain that are activated in response to disease-related emotional information, following whole lung allergen challenge in asthma. They propose that activity in these central nervous system locations, as measured by fMRI, is associated with the intensity of allergic inflammation, provoked by segmental bronchial challenge, in the absence of significant airflow obstruction. The investigators predict that this relationship will be mediated by changes in expression of genes in the IL-1β/IL-17 pathway.

DETAILED DESCRIPTION:
Asthma is characterized by airway inflammation, bronchial hyperresponsiveness and airflow obstruction. The development of symptoms in patients with asthma is initiated by exposure to a variety of airborne substances including aeroallergens. The inhalation of these allergens by asthmatic subjects initiates a series of complex, interactive immune events through activation of cell bound IgE, which serve to further existing airway inflammation, intensify underlying airway hyperresponsiveness and cause airflow obstruction. Although the immune events and processes associated with these reactions are largely localized to the airways themselves, a variety of other factors can contribute to the ongoing allergic response in either an enhancing or inhibitory manner. The regulation and modulation of these inflammatory actions is a key determinant to the eventual severity of asthma.

The initial step in the activation of the allergic airway response is the ability of inhaled allergen to activate IgE molecules on the pulmonary mast cell to release stored mediators and generate synthesis of new products, which can acutely contract airway smooth muscle. The mast cell also is capable of generating a variety of cytokines, which, in turn, can cause persistence and progression of the allergic response by furthering the underlying inflammation. In addition to mast cell activation, inhaled allergens are capable of stimulating resident lymphocytes in the lung. It is proposed that these allergen-responsive lymphocytes belong to a subpopulation of T helper cells (Th2), which are capable of generating a variety of cytokines, i.e. interleukin (IL)-4, IL-5, and IL-13. These Th2 cytokines can activate the local inflammatory response and can also serve to initiate events outside the lung, which can then further promote the persistence of the allergic inflammatory response.

To illustrate the means by which newly generated lung mediators can affect allergic inflammation, investigators have shown that inhaled allergen is associated with enhanced bone marrow generation of eosinophils. This enhanced bone marrow production of eosinophils is associated with bone marrow cell generation of IL-5, which causes terminal differentiation of eosinophils and their release into the circulation. Presumably, these recently generated eosinophils enter the circulation and are recruited to the lung where they may further the development of eosinophilic inflammation and the severity of asthma.

Other factors also influence the development and intensity of the allergic inflammatory response to inhaled allergen. In preliminary studies, the investigators have found that the stress associated with the final examination period in college students will enhance the eosinophilic inflammatory response to inhaled allergen. In addition, the investigators have found that during the final examination period, and independent of an allergen challenge, circulating eosinophils increase. Moreover, Marin and colleagues (2009) studied children with asthma over a two-year period and found that mononuclear cells from children who reported persistent life stress coupled with an acute stressful event produced elevated levels of asthma-promoting cytokines compared to asthmatic children without chronic stress or healthy controls. These findings suggest that the persistent stress associated with an acute stressor may promote allergic inflammatory events and that these processes include regulation of eosinophil numbers and recruitment to the lung.

From these studies, the investigators have evidence to suggest that stress-related events can influence allergic inflammation and, presumably, that these peripheral responses are regulated by central nervous system (CNS) events. Although stress-related events can modulate inflammatory processes, the mechanisms and CNS-site of this activity are poorly understood. It is proposed that areas of the brain are activated by stress and that these areas of activation may represent sites in the CNS that integrate information concerning the internal state of the body and signal the generation of modulating factors in the enhancement or inhibition of the allergic airway inflammation. To visualize these potential sites of CNS activation in asthma, it is possible to use neuroimaging techniques, such as positron emission tomography (PET) or functional magnetic resonance imaging (fMRI). The investigators have completed two prior studies that used fMRI to evaluate the central mechanisms associated with allergic inflammation, and in both studies, the anterior insula was identified as a region activated by asthma-related emotional cues that predicted the subsequent development of airway inflammation (e.g. Rosenkranz, M et al (2005) Proceedings of the National Academy of Science 102, 13319-13324.). In addition, the investigators have completed a study using PET to evaluate the neural mechanisms through which stress along contributes to asthma-related inflammation in individuals with high and low levels of chronic stress. This study corroborated our findings using fMRI, showing involvement of the insula, and also revealed new mechanisms involving IL-1β/IL-17 as a potential pathway linking through which stress-reactivity primes airway inflammation.

In the research described here, these two experimental paradigms will be merged to 1) determine the contribution of the IL-1β/IL-17 pathway in response of emotion neural circuitry provoked by airway inflammation in the absence of bronchoconstriction and 2) to determine the neural mechanisms and impact of acute stress on the airway inflammatory response to whole lung allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with no health concerns that might affect the outcome of the study,
* Physician diagnosis of asthma for at least six months prior to screening,
* FEV1 > or equal to 70% at baseline AND 12% reversibility OR PC20 response to methacholine < or equal to 16.0 mg/ml.
* Skin test positive to house dust mite (D. farinae), short ragweed or cat hair
* Asthma medications consisting of only inhaled short-acting B-agonist taken as needed,
* At least a 20% decrease in FEV1 during the immediate response following inhaled antigen challenge (historical data up to 5 years old will satisfy this criteria),
* Safety laboratory assessments within normal ranges (labs to include CBC with differential, PT, PTT and platelet count),
* Women of child-bearing potential (WCBP) must have a negative urine pregnancy test (urine HCG) within 48 hours of the methacholine challenge, within 48 hours of the inhaled allergen challenge and on the day of the segmental allergen challenge, as well as fMRI and PET scans. WCBP must agree to use a reliable method of birth control for the duration of the study (reliable methods of birth control can include abstinence, barrier methods, oral contraceptives, injection contraceptives or skin absorption contraceptives).
* In the opinion of the investigator, capable and willing to grant written informed consent and cooperate with study procedures and requirements.
* Ability to tolerate a simulated fMRI and PET brain scanning session, and
* Ability to give valid informed consent to participate by signing and dating a written consent form.

Exclusion Criteria:

* Psychotropic medication use that might affect function of neurocircuitry implicated in our hypotheses (at the discretion of the PI),
* Needle phobia or claustrophobia,
* Unable to distinguish colors used in Stroop task,
* Night shift work,
* Major health problems such as autoimmune disease, heart disease, type I and II diabetes, uncontrolled hypertension or lung diseases other than asthma. The listed health problems are definitive exclusion but decisions regarding major health problems not listed will be based upon the judgment of the investigator,
* History of a diagnosed Bipolar Disorder, Schizophrenia, or Schizoaffective Disorder,
* History of serious head trauma or seizure disorder (can be included at the discretion of the PI),
* No pre-existing chronic infectious disease,
* Any condition for which, in the opinion of the investigator, transient oxyhemoglobin desaturation is inadvisable,
* Pregnant or lactating females or has a planned pregnancy during the course of the study,
* Medication other than for asthma, allergies or contraception (at the discretion of the PI),
* Inhaled corticosteroids or oral corticosteroids within 1 month of screening,
* Upper or lower respiratory infection within 1 month of screening,
* Unstable asthma as indicated by self-report of increased symptoms or increased beta-agonist use over the 2 weeks preceding the screening visit,
* Currently receiving immunotherapy,
* Current smokers (defined as smoked within the last year) or a former smoker with a history of >5 pack years,
* Obesity as defined by a Body Mass Index (BMI) >35 or at the discretion of the principal investigator or co-investigator. Subjects with a BMI between 30 and 35 will be evaluated on a case by case basis by the PI or Co-I to determine eligibility.
* Use of an investigational drug within 30 days of entering the study. This criteria will be reviewed on a case by case basis by the principal investigator or co-investigator to determine appropriate washout period. Appropriate wash out period may be greater than 30 days depending on the half-life of the investigational drug,
* History of noncompliance with medical regiments or subjects who are considered unreliable including those with a psychiatric history that, in the opinion of the investigator, may interfere with the conduct of study procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with mild allergic asthma and across the full range of chronic stress levels will be recruited for study. Investigators will ensure this population includes participants in the top and bottom 10th percentiles of chronic stress.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Bronchoalveolar Eosinophils pre vs post antigen challenge | 48 hours
  The percent of eosinophils will be measured from the Bronchoalveolar lavage fluid pre segmental allergen challenge and will be measured 48 hours post segmental allergen challenge.

SECONDARY OUTCOMES:
Sputum Eosinophils pre stress condition vs post stress condition | 72 hours
  The percent of eosinophils will be measured from the sputum fluid pre stress condition and will be measured up to 72 hours later (post stress condition).
Sputum Eosinophils pre control condition vs post control condition | 72 hours
  The percent of eosinophils will be measured from the sputum fluid pre control condition and will be measured up to 72 hours later (post control condition).

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, MD, Principal Investigator — UW Madison
Locations (1):
- UW Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided